CLINICAL TRIAL: NCT03467594
Title: BE@Work: A Pilot Controlled Before and After Trial of a Workplace Physical Activity Programme.
Brief Title: BE@Work: Brief Exercise at Work
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Naomi Burn, PhD Researcher, Teesside University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 036/18
Record Dates: First submitted 2018-03-05; First posted 2018-03-16 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: High-intensity Interval Training
MeSH Terms: interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): 8 week workplace based exercise programme, 3 exercise sessions each week. Exercises will be conducted in an interval training format (60 second exercise bursts, followed by 75 seconds rest). The exercise bursts are designed to elicit ≥85% of participants age predicted maximum heart rate and will be tailored to each individuals fitness level and ability. Exercise sessions will be supervised and conducted in groups, with the option to request individual one-to-one sessions if preferred.
  Outcome measures assessed at baseline and follow-up (8 weeks)
  Interventions: Behavioral: High-intensity interval training
- Control (No Intervention): Outcome measures only at baseline at follow-up (8 weeks)

INTERVENTIONS:
Behavioral: High-intensity interval training — • Exercises will be conducted in an interval training format (60 second exercise bursts, followed by 75 seconds rest). The exercise bursts are designed to elicit ≥85% of participants age predicted maximum heart rate and will be tailored to each individuals fitness level and ability. Exercise sessions will be conducted 3 times per week for 8 weeks and will last between 15-25 minutes.
  Arms: Intervention arm

SUMMARY:
BE@Work (Brief Exercise at Work) is a pilot controlled before and after trial of a workplace physical activity programme.

DETAILED DESCRIPTION:
The aim of this study is to investigate the effect of an 8 week workplace physical activity programme on various markers of physical fitness, cardiometabolic health and wellbeing of employees. The primary outcome measures are the following: aerobic fitness, grip strength, leg extensor power, blood pressure, fasting blood glucose levels, lipid profiles, body mass index, waist and hip circumference and self-report measures of psychological wellbeing. The secondary outcome measure is total physical activity. The primary and secondary outcomes measures will be assessed in the control and intervention groups at baseline and at the end of the intervention (8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adult (≥18 years) with no health conditions that preclude them from exercise (information obtained via their self-report) and able to understand written and spoken English. Participants will be cleared for exercise participation via the Physical Activity Readiness Questionnaire Plus (PARQ+)

Exclusion Criteria:

* Exclusion criteria are: Individuals who are not cleared for exercise participation via the PARQ+ will not be eligible to participate. Additionally those unable or unwilling to give informed consent, have any diagnosis or symptoms of cardiovascular or metabolic disease (such as history of heart attack, stroke or diabetes), have been advised by a health professional to avoid physical exercise or activity, are pregnant or might be pregnant and cannot understand and speak English will not be eligible to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Aerobic fitness | 8 weeks
  Chester step test. This involves stepping onto and off a box at a height relevant to the participants age and usual physical activity level, at a set pace for a maximum of 10 minutes or until the participants heart rate reaches ≥80% of age-predicted maximum, whichever is first. Second-to-second heart rate (HR) will be monitored using a wrist worn heart rate monitor (Polar A360, Polar Electro Oy, Finland).
Alternative measure of aerobic fitness | 8 weeks
  If the participant chooses, they can also have their aerobic fitness measured using a ramp test. This will involve attending the Exercise Physiology Laboratory at Teesside University. Peak oxygen uptake will be measured by a ramp test on an electromechanically braked cycle ergometer (Lode Excalibure, Groningen, Netherlands). Participants will perform 5 minutes of submaximal exercise as a standard warm-up. Beginning with no load, power output will increase by 30 Watts (W) per minute until volitional exhaustion or the subject can no longer maintain a pedal cadence of 70-90 revolutions per minute. Expired gas will be collected and analysed throughout (Zan 600 USB CPX, nSpire Health Inc., United Kingdom), with peak oxygen uptake defined as the peak value of a 5-point average data set).
Hand grip strength | 8 weeks
  Hand grip strength will be measured using a hand dynamometer. The participant will stand with arms at their side, not touching their body holding the dynamometer in their non-dominant hand. The participant will be asked to squeeze the dynamometer with as much force as possible.
Leg extensor power | 8 weeks
  Leg extensor power will be assessed using the Nottingham leg extensor power rig, (Medical Engineering Unit, University of Nottingham, Nottingham, UK). The participant is seated in an adjustable seat and presses a foot pedal until the leg is extended. This petal accelerates a flywheel, and it is this average power in watts that is measured.
Resting blood pressure | 8 weeks
  Resting blood pressure will be measured using an electronic blood pressure monitor (Omron, M6 AC ME, Omron Healthcare, Kyoto, Japan).
Blood lipid concentration | 8 weeks
  Blood lipids will be assessed from a finger prick blood sample using the Cholestech LDX analyser (Cholestech Corporation, Hayward, CA, USA). The LDX analyser is currently used for the National Health Service Health Checks. Standard aspectic techniques will be used. A small puncture will be made in the middle finger using a one piece single use finger stick. The sample will be drawn into a 35 μL capillary tube and immediately transferred into a cassette sample well. The cassette will then be placed into the device drawer for analysis.
Body Mass Index | 8 weeks
  Body mass index will be calculated using the standard formula in units of kg/m2. Measurements of height and body mass will be taken using a standard scale and stadiometer.
Health related quality of life | 8 weeks
  Health related quality of life will be measured using a validated self-report paper based questionnaire (SF-36) (RAND, 2016). High scores mean higher quality of life.
Mental wellbeing | 8 weeks
  Mental wellbeing will be assessed using a validated self-report paper based questionnaire (Warwick Edinburgh Mental Wellbeing Scale) (Tennant et al., 2007). The total score is obtained by summing the score for each of the 14items. Total scores range from 14-70, higher scales indicate higher mental wellbeing.
Stress | 8 weeks
  Stress will be measured using a validated self-report paper based questionnaire (Perceived Stress Scale) (Cohen & Williamson, 1988). Scores ranging from 0-13, 14-26 and 27-40 would be considered low, medium and high perceived stress, respectively.
Blood glucose concentration | 8 weeks
  Fasting blood glucose (mmol/L) will be assessed from a finger prick blood sample using the Cholestech LDX analyser (Cholestech Corporation, Hayward, CA, USA). The LDX analyser is currently used for the National Health Service Health Checks. Standard aspectic techniques will be used. A small puncture will be made in the middle finger using a one piece single use finger stick. The sample will be drawn into a 35 μL capillary tube and immediately transferred into a cassette sample well. The cassette will then be placed into the device drawer for analysis.
Waist circumference | 8 weeks
  Waist and hip circumference will be measured using non-elastic Gulick tape measure (G-tape) at the narrowest point of the waist and broadest part of the hip.

SECONDARY OUTCOMES:
Accelerometer assessed habitual physical activity | 8 weeks
  Measurement of habitual physical activity over a 7 day period will be assessed using a Uniaxial Actigraph accelorometer (GT1M model, Actigraph, LLC, Pensacola, Florida). The participant will wear a small hip mounted accelerometer to assess their habitual physical activity for 7 days following their baseline data collection.

CONTACTS AND LOCATIONS:
Locations (1):
- Teesside University, Middlesbrough, United Kingdom

IPD SHARING:
Plan to Share IPD: No